CLINICAL TRIAL: NCT00827060
Title: Observation of the Initial Procalcitonin Values and the Clinical Course of Patients With Acute Respiratory Tract Infections at General Medical Practices in Greater Hannover
Brief Title: Observation of Initial Procalcitonin and the Clinical Course of Patients With Acute Respiratory Tract Infections
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Prof. Dr. med. Tobias Welte, Prof. Dr. med. Tobias Welte
Other Study IDs: HannoverPro
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Respiratory Tract Infections
Keywords: primary care; procalcitonin; acute respiratory tract infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Observation of the initial Procalcitonin values and the clinical course of consecutively included patients with Acute Respiratory Tract Infections at general medical practices in greater Hannover.

DETAILED DESCRIPTION:
Primary endpoint:

* initial Procalcitonin values of patients with Acute Respiratory Tract Infections

Secondary endpoints:

* correlation of initial Procalcitonin values to classify Acute Respiratory Tract Infections
* correlation of initial Procalcitonin values to subjective severity of Acute Respiratory Tract Infections
* correlation of initial Procalcitonin values to antibiotic- prescriptions
* correlation of initial Procalcitonin values to frequency of admission to hospital
* correlation of initial Procalcitonin values to frequency of referrals (radiology, pneumology)

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* all types of respiratory tract infection according to investigator´s diagnosis

Exclusion Criteria:

* pretreatment with antibiotics in the past 2 weeks
* portal hypertension
* Major surgeries or multiple trauma which require hospitalization, in previous 4 weeks
* Autoimmune disease and systemic diseases (lupus erythematodes, wegener´s disease)
* Peritoneal dialysis
* Acute treated or recently operated medullary c-cell-carcinoma, SCLC, carcinoid
* Other inflammatory diseases (e.g. urinary tract infection, pyelonephritis, pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care patients in 45 practices in greater Hannover
Sampling Method: Probability Sample
Enrollment: 702 (Actual)
Dates: Start 2006-12; Primary Completion 2007-06 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Burkhardt, PD Dr. med., Principal Investigator — Medical School Hannover
Locations (1):
- Medical School Hannover, Department Pneumology, Hanover, Germany

REFERENCES:
- [Derived] Burkhardt O, Ewig S, Haagen U, Giersdorf S, Hartmann O, Wegscheider K, Hummers-Pradier E, Welte T. Procalcitonin guidance and reduction of antibiotic use in acute respiratory tract infection. Eur Respir J. 2010 Sep;36(3):601-7. doi: 10.1183/09031936.00163309. Epub 2010 Feb 25. PMID 20185423